CLINICAL TRIAL: NCT01680159
Title: A Clinical Study of Increased Dose of TA-650 in Patients With Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-650-24
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis; Psoriatic Arthritis; Pustular Psoriasis (Excluding a Localized); Psoriatic Erythroderma
Keywords: Infliximab; REMICADE; TA-650; psoriasis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TA-650 (Experimental)
  Interventions: Drug: TA-650

INTERVENTIONS:
Drug: TA-650

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics of TA-650 at increased dose of 10 mg/kg every 8 weeks in patients with psoriasis in whom effect of the treatment was confirmed after the treatment with Remicade® at 5 mg/kg every 8 weeks but decreased thereafter.

DETAILED DESCRIPTION:
* Patients with plaque psoriasis or psoriatic arthritis:

  1. Screening Period:

     TA-650 at 5 mg per kg body weight is administered on the day of TA-650 administration at the start (week 0) and week 8 (if efficacy is not judged as decreased or maintained at week 8 of the screening period) , respectively, by intravenous infusion slowly over at least 2 hours.
  2. Increased Dose Period:

     If efficacy is judged as decreased in the screening period, TA-650 at 10 mg per kg body weight is administered on the day of TA-650 administration at the start (week 0) and at every 8 weeks up to week 32 in the increased dose period , respectively, as one dose by intravenous infusion slowly over at least 2 hours.
* Patients with pustular psoriasis or psoriatic erythroderma:

TA-650 at 10 mg per kg body weight is administered on the day of TA-650 administration at the start (week 0) and at every 8 weeks up to week 32, respectively, as one dose by intravenous infusion slowly over at least 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have already been diagnosed as having plaque psoriasis, psoriatic arthritis, pustular psoriasis (excluding a localized), or psoriatic erythroderma.
* Patients in whom effect of the treatment was confirmed for a certain period after the start of administration of Remicade® at 5 mg/kg at every 8 weeks but decreased thereafter.

Exclusion Criteria:

* Patients who have guttate psoriasis.
* Patients who have drug-induced psoriasis
* Patients who have previously used any other biological products than infliximab.
* Patients who have a concomitant diagnosis, or a history within 6 months prior to provisional enrollment, of serious infections that need hospitalization.
* Patients who have a concomitant diagnosis, or a history within 6 months prior to provisional enrollment, of opportunistic infections
* Female patients who are pregnant, breast-feeding, or possibly pregnant.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hideshi Torii, MD, Study Director — Social Insurance Central General Hospital; Kazuoki Kondo, MD, Study Director — Mitsubihsi Tanabe Pharma Corporation; Hidemi Nakagawa, MD, Study Chair — The Jikei University School of Medicine
Locations (7):
- Japan (7):
  - Investigational site, Chugoku
  - Investigational site, Chūbu
  - Investigational site, Hokkaido
  - Investigational site, Kanto
  - Investigational site, Kinki
  - Investigational site, Kyushu
  - Investigational site, Tōhoku

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients of Pustular Psoriasis and Psoriatic Erythroderma could directly receive doses of TA-650 10mg per 1kg not to go though screening period.
Groups:
- TA-650: During the normal dose period, patients received doses of TA-650 5 mg per 1 kg body weight as a slow intravenous infusion over at least 2 hours on the treatment day at week 0, and at week 8 (if patients were not assessed as being either "efficacy attenuated" or "efficacy maintained" at week 8 of the normal dose period).
Period: Screening Period
Arm/Group | TA-650
Started | 46
Completed | 39
Not Completed | 7
Not completed — Not meet criteria for dose-up period | 7
Period: Increased Dose Period
Arm/Group | TA-650
Started | 51
Completed | 43
Not Completed | 8
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Plaque Psoriasis; Psoriatic Arthritis; Pustular Psoriasis; Psoriatic Erythroderma: From week 0 to week 32, at 8-week intervals, patients received single doses of TA-650 10 mg per 1 kg body weight on each treatment day, as slow intravenous infusions administered over at least 2 hours.
- Total: Total of all reporting groups
Arm/Group | Plaque Psoriasis | Psoriatic Arthritis | Pustular Psoriasis | Psoriatic Erythroderma | Total
Number analyzed (Participants) | 31 | 8 | 7 | 5 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.9) | 50.1 (11.9) | 36.7 (9.7) | 55.8 (12.5) | 49.5 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 5 | 4 | 4 | 38
  Male | 6 | 3 | 3 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving 75% Improvement in the Psoriasis Area and Severity Index (PASI) Score
Description: The investigator or the subinvestigator examined the head, trunk, and upper and lower limbs, and assessed skin findings (erythema, induration, and scaling [scale]) at each of the regions and the extent of area affected. Total sores were calculated scores of the each regions.
  When the day of the assessment fell on a day on which study product was to be administered, the assessment was performed before the study product was administered.
  As a rule, the PASI score assessments for each patient were performed by the same investigator throughout the study, unless there was a special reason why this was not done (e.g., the investigator changed jobs).
  The number and percentage of patients achieving a 75% improvement in their PASI scores at each assessment time point.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 in Increased Dose Period
Measure: Number; unit: percentage of participants
Groups:
- Overall; Plaque Psoriasis; Psoriatic Arthritis; Pustular Psoriasis; Psoriatic Erythroderma: From week 0 to week 32, at 8-week intervals, patients received single doses of TA-650 10 mg per 1 kg body weight on each treatment day, as slow intravenous infusions administered over at least 2 hours.
Arm/Group | Overall | Plaque Psoriasis | Psoriatic Arthritis | Pustular Psoriasis | Psoriatic Erythroderma
Number analyzed (Participants) | 51 | 31 | 8 | 7 | 5
percentage of participants
  Week 0 (n=51,31,8,7,5) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 4 (n=51,31,8,7,5) | 13.7 | 16.1 | 0.0 | 0.0 | 40.0
  Week 8 (n=50,31,8,6,5) | 18.0 | 16.1 | 0.0 | 33.3 | 40.0
  Week 12 (n=49,30,8,6,5) | 36.7 | 40.0 | 0.0 | 50.0 | 60.0
  Week 16 (n=48,29,8,6,5) | 31.3 | 34.5 | 0.0 | 50.0 | 40.0
  Week 20 (n=46,28,7,6,5) | 50.0 | 53.6 | 14.3 | 50.0 | 80.0
  Week 24 (n=45,27,7,6,5) | 40.0 | 40.7 | 42.9 | 33.3 | 40.0
  Week 28 (n=44,26,7,6,5) | 63.6 | 69.2 | 28.6 | 83.3 | 60.0
  Week 32 (n=44,26,7,6,5) | 45.5 | 38.5 | 42.9 | 50.0 | 80.0
  Week 36 (n=44,26,7,6,5) | 47.7 | 42.3 | 28.6 | 66.7 | 80.0
  Week 40 (n=43,26,7,5,5) | 44.2 | 30.8 | 42.9 | 80.0 | 80.0

2. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score
Description: Score range is 0-72. Higher values represent a worse outcome. The investigator or the subinvestigator examined the head, trunk, and upper and lower limbs, and assessed skin findings (erythema, induration, and scaling [scale]) at each of the regions and the extent of area affected. Total sores were added scores of the each regions.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 in Increased Dose Period
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Overall | Plaque Psoriasis | Psoriatic Arthritis | Pustular Psoriasis | Psoriatic Erythroderma
Number analyzed (Participants) | 51 | 31 | 8 | 7 | 5
units on a scale
  Week 0 (n=51,31,8,7,5) | 14.70 [3.0 to 44.0] | 12.80 [4.6 to 44.0] | 13.95 [3.0 to 29.2] | 14.70 [3.1 to 37.2] | 22.20 [14.7 to 35.2]
  Week 4 (n=51,31,8,7,5) | 7.60 [0.6 to 30.7] | 6.20 [1.0 to 29.4] | 8.20 [0.6 to 28.0] | 9.90 [3.0 to 19.3] | 9.20 [4.2 to 30.7]
  Week 8 (n=50,31,8,6,5) | 7.25 [0.8 to 46.0] | 7.50 [1.0 to 46.0] | 8.20 [0.8 to 27.6] | 4.20 [1.2 to 34.8] | 14.00 [3.5 to 34.7]
  Week 12 (n=49,30,8,6,5) | 4.40 [0.7 to 39.3] | 4.40 [0.7 to 39.3] | 6.60 [0.8 to 24.1] | 3.70 [1.2 to 20.9] | 3.40 [1.6 to 25.7]
  Week 16 (n=48,29,8,6,5) | 6.80 [0.4 to 39.6] | 6.60 [0.4 to 16.2] | 6.60 [1.3 to 24.9] | 7.40 [0.4 to 23.0] | 9.50 [1.5 to 39.6]
  Week 20 (n=46,28,7,6,5) | 3.80 [0.0 to 22.0] | 3.95 [0.0 to 10.9] | 3.80 [1.2 to 22.0] | 4.80 [2.1 to 15.8] | 3.40 [1.2 to 14.8]
  Week 24 (n=45,27,7,6,5) | 4.80 [0.4 to 27.9] | 4.70 [0.4 to 15.1] | 4.80 [0.4 to 18.8] | 5.80 [2.0 to 14.0] | 5.60 [2.4 to 27.9]
  Week 28 (n=44,26,7,6,5) | 3.25 [0.0 to 20.4] | 3.25 [0.0 to 11.9] | 4.20 [0.0 to 20.4] | 2.75 [0.8 to 6.3] | 5.30 [0.9 to 11.6]
  Week 32 (n=44,26,7,6,5) | 4.70 [0.0 to 25.3] | 4.50 [0.0 to 21.6] | 4.20 [0.4 to 16.4] | 6.05 [1.2 to 8.8] | 4.80 [0.9 to 25.3]
  Week 36 (n=44,26,7,6,5) | 3.40 [0.0 to 29.8] | 3.40 [0.0 to 18.3] | 1.80 [0.0 to 29.8] | 3.15 [2.5 to 11.7] | 3.90 [0.9 to 24.6]
  Week 40 (n=43,26,7,5,5) | 3.70 [0.0 to 29.3] | 4.70 [0.0 to 27.6] | 2.40 [0.8 to 29.3] | 2.70 [2.1 to 6.2] | 3.30 [2.7 to 14.7]

3. Secondary Outcome: Percentage of Participants With Cleared and Minimal Skin Lesions of Physician Global Assessment (PGA) (Only for Patients With Plaque Psoriasis)
Description: The investigator or the subinvestigator made a global assessment of skin lesions in terms of the degree of erythema, induration, and scaling (scale), using the following 6-point scale (0 to 5). When the day of the assessment fell on a day on which study product was to be administered, the assessment was performed before the study product was administered. As a rule, the PGA for each patient were performed by the same investigator or subinvestigator throughout the study, unless there was a special reason why this was not done (e.g., the investigator or the subinvestigator changed jobs). Outcome measure data table is reported percentage of participants with Cleared and Minimal skin lesions.
  0: Cleared, 1: Minimal, 2: Mild, 3: Moderate, 4: Marked, 5: Severe
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 in Increased Dose Period
Measure: Number; unit: percentage of participants
Arm/Group | Plaque Psoriasis
Number analyzed (Participants) | 31
percentage of participants
  Week 0 (n=31) | 0.0
  Week 4 (n=31) | 32.3
  Week 8 (n=31) | 32.3
  Week 12 (n=30) | 43.3
  Week 16 (n=29) | 41.4
  Week 20 (n=28) | 57.1
  Week 24 (n=27) | 40.7
  Week 28 (n=26) | 69.2
  Week 32 (n=26) | 57.7
  Week 36 (n=26) | 61.5
  Week 40 (n=26) | 46.2

4. Secondary Outcome: Visual Analog Scale（VAS） of Pain Assessment by Subjects (Only for Patients With Psoriatic Arthritis)
Description: From 0 (best) to 100 (worst)
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 in Increased Dose Period
Measure: Median (Full Range); unit: mm
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 8
mm
  Week 0 (n=8) | 59.5 [10 to 92]
  Week 4 (n=8) | 19.0 [5 to 67]
  Week 8 (n=8) | 49.5 [4 to 98]
  Week 12 (n=8) | 14.0 [4 to 64]
  Week 16 (n=8) | 41.0 [5 to 96]
  Week 20 (n=7) | 27.0 [4 to 78]
  Week 24 (n=7) | 28.0 [4 to 72]
  Week 28 (n=7) | 17.0 [3 to 78]
  Week 32 (n=7) | 10.0 [6 to 80]
  Week 36 (n=7) | 8.0 [2 to 49]
  Week 40 (n=7) | 27.0 [2 to 64]

5. Secondary Outcome: Assessment of Severity (Only for Patients With Pustular Psoriasis)
Description: From 0 (best) to 17 (worst)
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 in Increased Dose Period
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Pustular Psoriasis
Number analyzed (Participants) | 7
units on a scale
  Week 0 (n=7) | 4.0 [4 to 10]
  Week 4 (n=7) | 3.0 [1 to 6]
  Week 8 (n=6) | 1.5 [1 to 10]
  Week 12 (n=6) | 1.5 [1 to 6]
  Week 16 (n=6) | 1.5 [1 to 9]
  Week 20 (n=6) | 2.0 [1 to 4]
  Week 24 (n=6) | 2.0 [1 to 5]
  Week 28 (n=6) | 1.0 [1 to 4]
  Week 32 (n=6) | 1.5 [1 to 4]
  Week 36 (n=6) | 1.0 [1 to 5]
  Week 40 (n=5) | 1.0 [1 to 4]

ADVERSE EVENTS:
Groups:
- TA-650（Normal Dose Period）Overall: Overall(Plaque Psoriasis・Psoriatic Arthritis)
- TA-650（Normal Dose Period）Plaque Psoriasis; TA-650（Dose Escalation Period）Plaque Psoriasis; TA-650（Entire Evaluation Period）Plaque Psoriasis: Plaque Psoriasis
- TA-650（Normal Dose Period）Psoriatic Arthritis; TA-650（Dose Escalation Period）Psoriatic Arthritis; TA-650（Entire Evaluation Period）Psoriatic Arthritis: Psoriatic Arthritis
- TA-650（Dose Escalation Period）Overall: Overall(Plaque Psoriasis・Psoriatic Arthritis・Pustular Psoriasis・Psoriatic Erythroderma)
- TA-650（Dose Escalation Period）Pustular Psoriasis: Pustular Psoriasis
- TA-650（Dose Escalation Period）Psoriatic Erythroderma: Psoriatic Erythroderma
Arm/Group | TA-650（Normal Dose Period）Overall | TA-650（Normal Dose Period）Plaque Psoriasis | TA-650（Normal Dose Period）Psoriatic Arthritis | TA-650（Dose Escalation Period）Overall | TA-650（Dose Escalation Period）Plaque Psoriasis | TA-650（Dose Escalation Period）Psoriatic Arthritis | TA-650（Dose Escalation Period）Pustular Psoriasis | TA-650（Dose Escalation Period）Psoriatic Erythroderma | TA-650（Entire Evaluation Period）Plaque Psoriasis | TA-650（Entire Evaluation Period）Psoriatic Arthritis
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/36 | 0/10 | 5/51 | 4/31 | 0/8 | 1/7 | 0/5 | 4/36 | 0/10
Other Adverse Events (participants affected / at risk) | 24/46 | 19/36 | 5/10 | 47/51 | 30/31 | 7/8 | 6/7 | 4/5 | 34/36 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650（Normal Dose Period）Overall (N=46) | TA-650（Normal Dose Period）Plaque Psoriasis (N=36) | TA-650（Normal Dose Period）Psoriatic Arthritis (N=10) | TA-650（Dose Escalation Period）Overall (N=51) | TA-650（Dose Escalation Period）Plaque Psoriasis (N=31) | TA-650（Dose Escalation Period）Psoriatic Arthritis (N=8) | TA-650（Dose Escalation Period）Pustular Psoriasis (N=7) | TA-650（Dose Escalation Period）Psoriatic Erythroderma (N=5) | TA-650（Entire Evaluation Period）Plaque Psoriasis (N=36) | TA-650（Entire Evaluation Period）Psoriatic Arthritis (N=10)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Bacterial pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650（Normal Dose Period）Overall (N=46) | TA-650（Normal Dose Period）Plaque Psoriasis (N=36) | TA-650（Normal Dose Period）Psoriatic Arthritis (N=10) | TA-650（Dose Escalation Period）Overall (N=51) | TA-650（Dose Escalation Period）Plaque Psoriasis (N=31) | TA-650（Dose Escalation Period）Psoriatic Arthritis (N=8) | TA-650（Dose Escalation Period）Pustular Psoriasis (N=7) | TA-650（Dose Escalation Period）Psoriatic Erythroderma (N=5) | TA-650（Entire Evaluation Period）Plaque Psoriasis (N=36) | TA-650（Entire Evaluation Period）Psoriatic Arthritis (N=10)
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 4 | 4 | 0 | 14 | 7 | 1 | 3 | 3 | 8 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 4 | 2 | 1 | 1 | 0 | 2 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 2 | 0 | 1 | 0 | 2 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 4 | 3 | 0 | 1 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Double stranded DNA antibody positive (Investigations) | 16 | 12 | 4 | 25 | 18 | 2 | 3 | 2 | 25 | 6
Interleukin level increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other